CLINICAL TRIAL: NCT07130695
Title: Olutasidenib Single Agent as Maintenance Therapy in IDH1mut AML After Induction and Consolidation
Brief Title: Olutasidenib Single Plus Combo Therapy in IDH1mut AML After Induction and Consolidation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-25-22096
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olutasidenib Investigational Agent Administration (Experimental): 150 mg by mouth twice daily.
  Interventions: Drug: Olutasidenib Investigational Agent Administration

INTERVENTIONS:
Drug: Olutasidenib Investigational Agent Administration — Twice daily olutasidenib maintenance therapy

SUMMARY:
Treatment with olutasidenib for isocitrate dehydrogenase 1 (IDH1) mutant acute myeloid leukemia (AML) after completion of traditional intensive induction/consolidation is likely to be safe, tolerable, and may provide clinical benefit in terms of maintenance of remission and perhaps improvement in survival.

DETAILED DESCRIPTION:
Up to 15 participants will receive treatment with olutasidenib 150 mg by mouth twice daily for up to 2 years. Participants will be regularly monitored for toxicities, adverse events, quality of life (QOL), and disease status. Once off treatment, participants will continue to be followed for a maximum of 2 years from date of enrollment for survival endpoints

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-acute promyelocytic isocitrate dehydrogenase (1 IDH1) mutant acute myeloid leukemia (AML). IDH1 mutation may be identified by NGS or PCR based methods and identified at time of diagnosis or any other time point prior to enrollment.
* Completed induction and/or consolidation intended as per treating physician to reach complete response (CR),complete response with partial hematologic recovery (CRh), or complete response with incomplete hematologic recovery (CRi), or morphologic leukemia free state (MLFS) at time of study enrollment Patients must be within 90 days of their last cycle of upfront therapy.
* Age ≥18 years
* Calculated creatinine clearance (by Cockroft-Gault) ≥30 mL/min
* Total bilirubin ≤2 × upper limit of normal (ULN) Note: patients with Gilbert's syndrome may be included if total bilirubin is ≤3 × ULN and direct bilirubin is ≤2 × ULN
* Serum aspartate aminotransferase/ alanine aminotransferase (AST/ALT) ≤3 × ULN
* Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2 or KPS >50%
* Able to take oral medications
* Women of childbearing potential must consent to effective contraception during study treatment and at least 6 months following the last dose. Effective methods of contraception include oral or injectable hormonal birth control, intrauterine device (IUD), and double- barrier methods. (ie, combination of male condom with either cap, diaphragm or sponge with spermicide)
* Male participants who are sexually active with a woman of childbearing potential and who have not had vasectomies must be willing to use a barrier method of contraception and refrain from sperm donation from initial study drug until 90 days after last dose of study drug.

Exclusion Criteria:

* History of hypersensitivity or allergic reaction to olutasidenib or its components
* Corrected Q-T interval (QTc) (Fredericia calculation) > 450 ms (after corrective action is taken)
* History of Torsades de Pointes
* Any gastrointestinal condition thought by the treating investigator to impair oral absorption of medication
* Stem cell transplant eligible and planned within 60 days of study start date in the opinion of the treating investigator
* Uncontrolled intercurrent illness or infection (those with controlled human immunodeficiency virus (HIV), hepatitis, or other chronic infections are eligible)
* Female participants who are pregnant or intend to donate eggs during the study or for 6 months after receiving their last dose of study drug
* Nursing women, women of childbearing potential with positive pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception. (Appropriate method(s) of contraception include oral or injectable hormonal birth control, IUD, and double-barrier methods)
* Male participants who intend to donate sperm during the course of this study or for 3 months after last dose
* Participants receiving, or are expected to require during the study, any concomitant medications that may interfere with efficacy, metabolism, or safety of the investigational agent, including drugs known to cause QT prolongation. for which drug interactions with olutasidenib would be prohibitory
* Concurrent chemotherapy for non-AML malignancy that is expected to interfere with the efficacy, metabolism, or safety of the agent under investigation
* Received non-intensive upfront therapy including hypomethylating agents (HMA) /Venetoclax based
* Currently receiving other targeted therapies or AML directed therapies, including but not limited to other IDH1 or IDH2 inhibitors, FMS-like tyrosine kinase 3 (FLT3) inhibitors, B-cell lymphoma 2 (BCL-2) inhibitors, menin inhibitors
* Other investigational agents in another clinical trial within 4 weeks prior to enrollment
* Systemic corticosteroids above physiologic replacement doses (10mg/day prednisone or equivalent), unless used to tread IDH differentiation syndrome or as part of a pre-specified protocol exception
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the participant's risk or limit the participant's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of olutasidenib after upfront acute myeloid leukemia (AML) therapy with intensive induction and/or consolidation in IDH1 mutant AML. | Up to 2 years
  Feasibility defined as the number of participants with 75% protocol treatment compliance for a duration of at least 4 cycles (to include protocol defined dose delays), or until disease relapse or allogeneic hematopoietic stem cell transplant (alloHCT).
Assess the tolerability of olutasidenib after upfront AML therapy with intensive induction and/or consolidation in IDH1 mutant AML | Up to 2 years
  Incidence of grade ≥4 adverse events (AEs) attributable to study drug for duration of treatment on study

SECONDARY OUTCOMES:
Measure progression free survival | Up to 2 years following end of treatment
  Progression free survival (PFS), defined as the time from the date of the first dose of study treatment to the date of relapse or death
Estimate overall survival (OS) | Up to 2 years following end of treatment
  Overall survival defined as the time from the date of diagnosis to the date of death.
Assess mean residual disease (MRD) negativity rates by both PCR based and flow cytometric methodologies | Baseline, Cycle 3 Day 15, and End of Treatment (Each cycle is 28 days)
  MRD status by multi-parameter flow cytometry at 10-5 sensitivity, by PCR based IDH1 sequencing assay, or by both methods of detection.
Estimate rates of ability to proceed with transplant given maintenance opportunities. | Up to 2 years
  Incidence of study patients receiving allogeneic hematopoietic stem cell transplant (alloHCT) within 2 years of initiating olutasidenib maintenance therapy.
Characterize quality of life (QOL) metrics by SF 36 | Cycle 1Day 1, Cycle 2 Day 1, Cycle 4 day 1, and End of Treatment (EOT) (Each cycle is 28 days)
  Health-related quality of life (HRQOL) metrics as assessed by Short Form (SF-36), a 36-item, patient-reported survey that assesses health-related quality of life. This survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The RAND-36 Health Survey is scored by first recoding the answers to a 0-100 scale, with higher scores indicating better health. (https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html)

CONTACTS AND LOCATIONS:
Overall Officials: Keri Maher, DO, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share individual patient data (IPD).